CLINICAL TRIAL: NCT07153848
Title: A Multicenter Cohort Study for Early Alzheimer's Disease in Zhejiang: an Observational Study on Lecanemab Treatment
Brief Title: An Observational Study on Lecanemab Treatment for Early Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: lecanamab and biomarkers
Record Dates: First submitted 2025-05-07; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
Keywords: lecanemab; Alzheimer Disease; biomarkers; blood
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- donepezil treatment: In this cohort, a standardized treatment regimen of donepezil at a dose of 10 mg was employed.
- donepezil and lencanemab treatment: The group was treated with a combination regimen of lencanumab and donepezil. Lencanumab was administered at a dose of 10 mg/kg every two weeks, while donepezil was used at a dose of 10 mg per day.

SUMMARY:
The goal of this observational study is to valuate the sensitivity and specificity of different blood biomarkers for monitoring and assessing Aβ-PET-confirmed mitigation of amyloid pathology by lencanumab treatment in subjects treated with lencanumab.

DETAILED DESCRIPTION:
This study was a prospective observational study of a patient population treated or planning to be treated with lencanemab from a multicenter cohort of patients with early-stage AD in Zhejiang Province. It was a real-world study based on the treatment of lencanemab. The primary enrollment population was patients with mild AD or mild AD-origin cognitive disorders who had completed positive Aβ-PET scans that met the PET quality-control criteria and who were receiving treatment with lencanemab. Patients with cognitive impairment were divided into two subgroups: those receiving donepezil treatment alone and those receiving lencanemab combined with standard treatment with donepezil. Fresh plasma was collected at baseline, 3 months of follow-up, 6 months of follow-up, 12 months of follow-up, and 18 months of follow-up, respectively. Amyloid PET scanning was performed at 12 months of follow-up and 18 months of follow-up. In order to evaluate the sensitivity and specificity of different blood biomarkers for monitoring and assessing the alleviation of amyloid pathology progression by Aβ-PET-confirmed lencanumab treatment, blinded peripheral blood AD core marker assays were performed in the main central laboratory. Furthermore, the aim was to provide a follow-up tool suitable for clinical blood marker-based monitoring of lencanumab treatment.

ELIGIBILITY:
Inclusion criteria (all of the following must be met simultaneously):

Mild Alzheimer's Disease (AD):

1. Age ≥ 45 years but ≤ 85 years;
2. Literacy level of elementary school and above (i.e., ≥3 years of education);
3. Fulfillment of the diagnostic criteria for probable AD in the NINCDS-ADRDA 2007 revision (or the diagnostic criteria for clinically probable AD in the National Institute on Aging and Alzheimer's Disease Association NIA-AA 2011 edition);
4. Clinical Dementia Rating Scale CDR-global = 1 point;
5. Aβ-PET scan suggesting extensive deposition of Aβ plaques in the brain.

AD-derived mild cognitive impairment (aMCI) inclusion criteria (must meet all of the following conditions at the same time):

1. Age: 45 years or older but ≤85 years;
2. Literacy level elementary school and above (i.e., ≥3 years of education);
3. Meeting Peterson's 2004 diagnostic criteria for MCI:

   (i) Complaint of memory impairment that can be confirmed by an informed person; (ii) objective evidence of memory impairment (memory test scores 1-1.5 standard deviations below normal controls matched for age and literacy; e.g., Huashan Hospital's recommended cut-off values for those with elementary school literacy or above are as follows: long-delayed recall 50-59 years old ≤ 5, 60-69 years old ≤ 4, 70-79 years old ≤ 3, 80-89 years old ≤ 2, or re-recognition scores of 50-59 years old ≤ 20, 60-69 age ≤19 points, 70-79 years ≤18 points, 80-89 years ≤16 points); (iii) Overall cognitive functioning was largely preserved, with CDR-global = 0.5 points and MMSE: ≥24 points for those with junior high school or higher education used in this study;

   ④ Daily life ability remains normal (basically able to complete going out by transportation and shopping and counting, etc.);

   ⑤ Does not meet the International Classification of Diseases Diagnostic Manual, 10th edition dementia criteria (for research purposes) and the National Institute of Neurological and Speech-Language Disorders and Stroke, Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) likely diagnostic criteria for AD dementia; (vi) Aβ-PET scan suggested extensive deposition of Aβ plaques in the brain.

Normal control Inclusion criteria (all of the following must be met simultaneously).

1. Age ≥55 years but ≤85 years;
2. Elementary school 3 years of education and above;
3. MMSE: ≥26 points for those with junior high school or higher education;
4. CDR=0;
5. Activity of Daily Living Scale (ADL) score ≤ 20;
6. No significant deposition of Abeta in the brain as indicated by Aβ-PET scan.

Exclusion Criteria (excluded if any of the following conditions were met):

1. Those with a history of stroke and neurologic focal signs, head MRI scans excluding external infarct foci, brain softening foci and other occupying lesions, etc., as well as SWI sequences showing 5 or more microhemorrhagic foci, vascular malformations, etc;
2. Presence of other neurological disorders that may cause brain dysfunction (e.g., schizophrenia, severe anxiety and depression, frontotemporal lobe dementia, Huntington's disease, brain tumors, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, traumatic brain injury, and normal cranial pressure hydrocephalus, etc.);
3. Presence of other systemic diseases that can cause cognitive impairment, such as hypothyroidism, folic acid and vitamin B12 deficiency, specific infections (e.g., syphilis, HIV), alcohol and drug abuse;
4. Presence of a history of severe hepatic or renal insufficiency, severe pulmonary insufficiency, severe anemia, severe gastrointestinal disorders, severe cardiac arrhythmias, cardiac infarction within 6 months, and malignant tumors;
5. Oral anticoagulants (including warfarin and new oral anticoagulants, etc.);
6. Presence of contraindications to NMR such as metal implantation in the body;
7. Diseases such as aphasia, impaired consciousness, etc. that prevent cooperation in completing the cognitive examination;
8. Refusal to sign the informed consent.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples from a multicenter study cohort of early AD in Zhejiang Province (real-world study based on lencanumab treatment)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with blood biomarkers | Fresh plasma was collected at baseline, 3 months of follow-up, 6 months of follow-up, 12 months of follow-up, and 18 months of follow-up, respectively
  Blinded peripheral blood AD core marker testing including but not limited to Aβ40, Aβ42, total tau, p-tau181/217, NFL, GFAP

SECONDARY OUTCOMES:
Aβ-PET | Amyloid PET scan at 12 months follow-up, 18 months follow-up
  Aβ-PET scanning was conducted on enrolled patients to evaluate alterations in the quantity of amyloid plaque deposits within their brains.
Cognitive funtion - MMSE | was collected at baseline, 3 months of follow-up, 6 months of follow-up, 12 months of follow-up, and 18 months of follow-up, respectively
  Multidimensional neuropsychological assessment is mainly used to assess the cognitive function of patients. MMSE is widely used in cognitive dysfunction which consists of the following ten parts: orientation, memory, attention and numeracy, ability to recall, language skills, including naming ability, retelling ability, three-step command, reading ability, writing ability. The values range from 0 to 30, with higher score indicating better outcome.
Cognitive funtion - MoCA | was collected at baseline, 3 months of follow-up, 6 months of follow-up, 12 months of follow-up, and 18 months of follow-up, respectively
  Multidimensional neuropsychological assessment is mainly used to assess the cognitive function of patients. MoCA is also an assessment tool for rapid screening of cognitive dysfunction, including 8 cognitive domains such as visual structure skills, executive function, memory, language, attention and concentration, calculation, abstract thinking and orientation. The values range from 0 to 30, with higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No